CLINICAL TRIAL: NCT04258020
Title: Exploratory Trial to Improve Postextubation Management for Patients at Risk for Extubation Failure
Brief Title: Postextubation Management in Patients at Risk for Extubation Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Significant impact of COVID pandemic on ability to conduct study
Sponsor: OhioHealth (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1332767
Record Dates: First submitted 2020-01-27; First posted 2020-02-06 (Actual); Results first posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Ventilatory Failure
MeSH Terms: conditions — Hypoventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental: alternating BiPAP and HFNC (Experimental): Patients will be placed on alternating BiPAP and HFNC for 24 hours following extubation
  Interventions: Device: BiPAP; Device: HFNC
- Historical Control: standard of care (No Intervention): A historical control cohort will be composed of patients treated according to their physician's standard of care following removal from mechanical ventilation.

INTERVENTIONS:
Device: BiPAP — Bilevel Positive Airway Pressure (BiPAP) oxygen administration
  Arms: Experimental: alternating BiPAP and HFNC
Device: HFNC — Heated High Flow Nasal Cannula oxygen administration
  Arms: Experimental: alternating BiPAP and HFNC

SUMMARY:
At the time of weaning from mechanical ventilation, patients with heart and/or lung conditions will be given oxygen support with alternating bilevel positive airway pressure (BiPAP; oxygen via face mask) and heated high flow nasal cannula oxygen (HFNC; oxygen via nasal cannula) to see if this method reduces the likelihood of re-intubation.

DETAILED DESCRIPTION:
It is clinically challenging to predict when patients can be successfully removed from mechanical ventilation (MV). Liberating high-risk patients such as the elderly and those with complex, chronic cardiac or pulmonary diseases from MV is particularly challenging.

Evidence from randomized trials and meta-analyses suggests that the type of postextubation supportive care provided, such as oxygen delivery via nose or mouth, may affect the risk of reintubation. However, it is unclear which of many possible postextubation management protocols results in the best patient outcomes, particularly for this subset of high-risk patients.

The purpose of this study is therefore to assess a standardized combined protocol of postextubation oxygen delivery consisting of early, alternating BiPAP with HFNC over 24 hours following extubation. BiPAP and HFNC are both currently provided to patients as standard of care, based on clinician judgement; however, the timing and nature of the methods are variable.

ELIGIBILITY:
Inclusion Criteria:

* Documented high-risk factors of interest [congestive heart failure (CHF), chronic obstructive pulmonary disease (COPD), and/or positive fluid balance]
* The modified rapid shallow breathing index on day of extubation must be between 58-105 breaths per minute per liter (breaths/min/L)
* Patient must successfully complete spontaneous breathing trial and be determined eligible for extubation
* Only primary extubations will be included

Exclusion Criteria:

* Undergoing terminal extubation or placed on comfort care
* Home ventilator use
* Any contraindication that would preclude the postextubation protocol (e.g., facial trauma, tracheotomy, or any other reason that would preclude use of BiPAP or HFNC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Devulapally, MD, Principal Investigator — OhioHealth
Locations (1):
- OhioHealth Grant Medical Center, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants in the experimental group withdrew from the study prior to intervention. One participant in the experimental group withdrew consent at time of regained capacity. Because the study was terminated (halted prematurely) no data were collected for the historical control group.
Period: Overall Study
Arm/Group | Experimental: Alternating BiPAP and HFNC | Historical Control: Standard of Care
Started | 4 | 0
Completed | 3 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Because the prospective group was terminated, no data collection for the historical control was collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Alternating BiPAP and HFNC | Historical Control: Standard of Care | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 2 |  | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 2 |  | 2
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Re-intubation Within 72 Hours
Description: The number of patients who require re-intubation
Time Frame: 72 hours following extubation
Population: Because the study was terminated (halted prematurely), no historical control data were collected
Measure: Number; unit: participants
Arm/Group | Experimental: Alternating BiPAP and HFNC | Historical Control: Standard of Care
Number analyzed (Participants) | 3 | 0
participants | 0 |

2. Secondary Outcome: Re-intubation Within 1 Week
Description: The number of patients who require re-intubation
Time Frame: 1 week following extubation
Population: Because the study was terminated (halted prematurely), no historical control data were collected
Measure: Number; unit: participants
Arm/Group | Experimental: Alternating BiPAP and HFNC | Historical Control: Standard of Care
Number analyzed (Participants) | 3 | 0
participants | 0 |

3. Secondary Outcome: Length of Stay
Description: Hospital length of stay
Time Frame: Through hospital discharge, an average of 10.9 ± 1.91 days
Population: Because the study was terminated (halted prematurely), no historical control data were collected
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Experimental: Alternating BiPAP and HFNC | Historical Control: Standard of Care
Number analyzed (Participants) | 3 | 0
Days | 10.9 (1.91) |

4. Secondary Outcome: Ventilator Time
Description: The total duration of time patients spend on a ventilator
Time Frame: Through hospital discharge, an average of 10.9 ± 1.91 days
Population: Because the study was terminated (halted prematurely), no historical control data were collected
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Experimental: Alternating BiPAP and HFNC | Historical Control: Standard of Care
Number analyzed (Participants) | 3 | 0
Days | 3.5 (1.33) |

5. Secondary Outcome: Mortality
Description: The proportion of patients who expire during the hospital stay
Time Frame: Through hospital discharge, an average of 10.9 ± 1.91 days
Population: Because the study was terminated (halted prematurely), no historical control data were collected
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Alternating BiPAP and HFNC | Historical Control: Standard of Care
Number analyzed (Participants) | 3 | 0
Participants | 0 |

6. Secondary Outcome: Adverse Event Rate
Description: The proportion of patients experiencing an adverse event
Time Frame: Through 1 week following extubation
Population: Because the study was terminated (halted prematurely), no historical control data were collected
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Alternating BiPAP and HFNC | Historical Control: Standard of Care
Number analyzed (Participants) | 3 | 0
Participants | 1 |

7. Secondary Outcome: 30-day Readmission
Description: The proportion of patients who require re-admission within 30 days of discharge
Time Frame: 30 days following discharge
Population: Because the study was terminated (halted prematurely), no historical control data were collected
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Alternating BiPAP and HFNC | Historical Control: Standard of Care
Number analyzed (Participants) | 3 | 0
Participants | 0 |

ADVERSE EVENTS:
Time Frame: Through hospital discharge, and average of 10.9 days.
Description: All patients were assessed for adverse events through hospital discharge
Arm/Group | Experimental: Alternating BiPAP and HFNC | Historical Control: Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 1/3 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Alternating BiPAP and HFNC (N=3) | Historical Control: Standard of Care (N=0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT04258020/Prot_SAP_001.pdf
  • Informed Consent Form (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT04258020/ICF_002.pdf